CLINICAL TRIAL: NCT04091061
Title: A PHASE 1, NON-RANDOMIZED, OPEN-LABEL, SINGLE-DOSE, PARALLEL-COHORT STUDY TO COMPARE THE PHARMACOKINETICS OF PF 06865571 IN ADULT PARTICIPANTS WITH VARYING DEGREES OF HEPATIC IMPAIRMENT RELATIVE TO PARTICIPANTS WITHOUT HEPATIC IMPAIRMENT
Brief Title: Effect Of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of PF-06865571 In Subjects With Hepatic Impairment and in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C2541009
Record Dates: First submitted 2019-09-13; First posted 2019-09-16 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Hepatic Impairment; Healthy Volunteers
Keywords: Non-alcoholic Fatty Liver Disease; Non-alcoholic steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ervogastat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PF-06865571 Moderate Hepatic Impairment (Experimental): This arm includes participants with moderate hepatic impairment who will receive an oral dose of PF-06865571 100 mg on Day 1
  Interventions: Drug: PF-06865571 100 mg
- PF-06865571 Severe Hepatic Impairment (Experimental): This arm includes participants with severe hepatic impairment who will receive an oral dose of PF-06865571 100 mg on Day 1
  Interventions: Drug: PF-06865571 100 mg
- PF-06865571 Mild Hepatic Impairment (Experimental): This arm includes participants with mild hepatic impairment who will receive an oral dose of PF-06865571 100 mg on Day 1
  Interventions: Drug: PF-06865571 100 mg
- PF-06865571 Healthy Participants (Experimental): This arm includes healthy participants who will receive an oral dose of PF-06865571 100 mg on Day 1
  Interventions: Drug: PF-06865571 100 mg

INTERVENTIONS:
Drug: PF-06865571 100 mg — PF-06865571 in 100 mg oral tablet will be administered on Day 1

SUMMARY:
The current study is proposed to evaluate whether there is any clinically meaningful effect of hepatic impairment on the plasma PK of PF-06865571.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Body mass index (BMI) of 17.5 to 35.4 kg/m2, inclusive; and a total body weight >50 kg (110 lb), at the Screening visit; with a single repeat assessment of total body weight (and hence BMI), on a separate day permitted to assess eligibility, if needed.
* Capable of giving signed informed consent.

Exclusion Criteria

* Any condition possibly affecting drug absorption (eg, prior bariatric surgery,gastrectomy, ileal resection).
* At Screening, participants with a positive result for human immunodeficiency virus (HIV) antibodies, as assessed by sponsor-identified central laboratory, with a single repeat permitted to assess eligibility, if needed.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study.
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of investigational product used in this study (whichever is longer).
* Participants with known prior participation (ie, randomized and received at least 1 dose of investigational product) in a study involving PF-06865571.
* A positive urine drug test, for illicit drugs on Day -1,
* At Screening or Day -1, a positive breath alcohol test.
* Male participants with partners who are currently pregnant.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing and until the follow-up contact.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-04-07 (Actual); Study Completion 2020-04-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - University of Miami Division of Clinical Pharmacology, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C2541009

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 32 participants screened for entry into the study, 24 participants were assigned and received a single, oral 100 mg dose of PF-06865571: 6 participants in each of the 4 hepatic function cohorts.
Groups:
- Cohort 1 (Without Hepatic Impairment): Hepatic function was categorized based on Child Pugh Score.
  NA for participants without hepatic impairment.
- Cohort 2 (Mild Hepatic Impairment): Hepatic function was categorized based on Child Pugh Score.
  Class A (5 to 6 points) for participants with mild hepatic impairment.
- Cohort 3 (Moderate Hepatic Impairment): Hepatic function was categorized based on Child Pugh Score.
  Class B (7 to 9 points) for participants with moderate hepatic impairment.
- Cohort 4 (Severe Hepatic Impairment): Hepatic function was categorized based on Child Pugh Score.
  Class C (10 to 15 points) for participants with severe hepatic impairment.
Period: Overall Study
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (3.92) | 58.2 (5.15) | 64.5 (5.32) | 57.5 (8.60) | 60.3 (6.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 0 | 3 | 10
  Male | 2 | 3 | 6 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 3 | 14
  Not Hispanic or Latino | 2 | 2 | 3 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 6 | 6 | 6 | 4 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax of PF-06865571 was observed directly from data.
Time Frame: For Cohort 1, pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48 hours post dose. For Cohorts 2-4, pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 16, 24, 36, 48, 72 hours post dose.
Population: All participants who received PF-06865571 and in whom at least 1 plasma concentration value was reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL) | 532.2 (153) | 835.5 (39) | 668.3 (35) | 658.6 (42)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other — 90% Confidence Intervals (CIs) for the ratios of adjusted geometric means (Test/Reference): Analysis 1: Mild Hepatic Impairment = Test, Without Hepatic Impairment = Reference; Ratio (%) = 156.99, 90% CI 2-sided [83.14 to 296.44] — 90% CIs for the ratios of adjusted geometric means (Test/Reference): Analysis 1: Mild Hepatic Impairment = Test, Without Hepatic Impairment = Reference
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other — 90% CIs for the ratios of adjusted geometric means (Test/Reference): Analysis 2: Moderate Hepatic Impairment = Test, Without Hepatic Impairment = Reference; Ratio (%) = 125.58, 90% CI 2-sided [66.51 to 237.13] — 90% CIs for the ratios of adjusted geometric means (Test/Reference): Analysis 2: Moderate Hepatic Impairment = Test, Without Hepatic Impairment = Reference
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other — 90% CIs for the ratios of adjusted geometric means (Test/Reference): Analysis 3: Severe Hepatic Impairment = Test, Without Hepatic Impairment = Reference; Ratio (%) = 123.75, 90% CI 2-sided [65.54 to 233.68] — 90% CIs for the ratios of adjusted geometric means (Test/Reference): Analysis 3: Severe Hepatic Impairment = Test, Without Hepatic Impairment = Reference

2. Primary Outcome: Area Under the Curve From Time 0 to Last Quantifiable Concentration (AUClast)
Description: AUClast of PF-06865571 was determined by linear/log trapezoidal method.
Time Frame: as for outcome 1
Population: All participants dosed who had at least 1 of the PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram*hour per milliliter (ng*hr/mL) | 2078 (155) | 3247 (40) | 3443 (42) | 3163 (47)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other — 90% CIs for the ratios of adjusted geometric means (Test/Reference): Analysis 1: Mild Hepatic Impairment = Test, Without Hepatic Impairment = Reference; Ratio (%) = 156.25, 90% CI 2-sided [81.07 to 301.16] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) = 165.66, 90% CI 2-sided [85.95 to 319.29] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other — [test comment as in outcome 1, analysis 3]; Ratio (%) = 152.18, 90% CI 2-sided [78.96 to 293.32] — [estimate comment as in outcome 1, analysis 3]

3. Primary Outcome: Area Under the Curve From Time 0 to Extrapolated Infinite Time (AUCinf)
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time 0 (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: as for outcome 1
Population: All participants dosed who had at least 1 of the PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 2083 (155) | 3250 (39) | 3445 (42) | 3171 (47)
Statistical Analysis 1: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 2 (Mild Hepatic Impairment); Test type: Other — [test comment as in outcome 2, analysis 1]; Ratio (%) = 156.00, 90% CI 2-sided [80.95 to 300.60] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 3 (Moderate Hepatic Impairment); Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) = 165.38, 90% CI 2-sided [85.82 to 318.67] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Cohort 1 (Without Hepatic Impairment) vs Cohort 4 (Severe Hepatic Impairment); Test type: Other — [test comment as in outcome 1, analysis 3]; Ratio (%) = 152.20, 90% CI 2-sided [78.99 to 293.29] — [estimate comment as in outcome 1, analysis 3]

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who receives study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs were events following start of treatment.
Time Frame: Up to Day 32 (31 days after investigational product administration)
Population: All participants who received PF-06865571.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities
Description: The following parameters were analyzed for laboratory examination: hematology, clinical chemistry, and urinalysis. The abnormalities with at least 1 participant are presented here.
Time Frame: Up to Day 4 (3 days after investigational product administration)
Population: All participants who received PF-06865571.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Hemoglobin <0.8xLower limit of normal (LLN) | 0 | 0 | 0 | 1
  Hematocrit <0.8xLLN | 0 | 0 | 0 | 1
  Erythrocytes (Ery.) <0.8xLLN | 0 | 0 | 0 | 1
  Ery. Mean Corpuscular Volume <0.9xLLN | 0 | 1 | 0 | 0
  Ery. Mean Corpuscular Volume >1.1xupper limit of normal (ULN) | 0 | 0 | 0 | 1
  Ery. Mean Corpuscular Hemoglobin <0.9xLLN | 0 | 1 | 0 | 0
  Ery. Mean Corpuscular Hemoglobin >1.1xULN | 0 | 0 | 0 | 2
  Platelets <0.5xLLN | 0 | 0 | 0 | 1
  Leukocytes <0.6xLLN | 0 | 0 | 0 | 1
  Lymphocytes <0.8xLLN | 0 | 0 | 0 | 1
  Neutrophils <0.8xLLN | 0 | 0 | 1 | 0
  Monocytes >1.2xULN | 0 | 0 | 1 | 0
  Activated Partial Thromboplastin Time >1.1xULN | 1 | 1 | 2 | 2
  Prothrombin Time >1.1xULN | 0 | 0 | 0 | 3
  Prothrombin International. Normalized Ratio >1.1xULN | 0 | 0 | 0 | 3
  Bilirubin >1.5xULN | 0 | 0 | 1 | 4
  Direct Bilirubin >1.5xULN: number analyzed (Participants) | 0 | 0 | 2 | 4
  Direct Bilirubin >1.5xULN | 0 | 0 | 1 | 4
  Indirect Bilirubin >1.5xULN: number analyzed (Participants) | 0 | 0 | 2 | 4
  Indirect Bilirubin >1.5xULN | 0 | 0 | 0 | 1
  Aspartate Aminotransferase >3.0xULN | 0 | 0 | 1 | 0
  Alanine Aminotransferase >3.0xULN | 0 | 0 | 1 | 0
  Gamma Glutamyl Transferase >3.0xULN | 0 | 0 | 0 | 1
  Albumin <0.8xLLN | 0 | 0 | 1 | 1
  Glucose >1.5xULN | 0 | 2 | 1 | 0
  Urine Glucose ≥1 | 0 | 0 | 0 | 1
  Urine Ketones ≥1 | 0 | 0 | 1 | 0
  Urine Protein ≥1 | 0 | 0 | 0 | 1
  Urine Hemoglobin ≥1 | 2 | 1 | 2 | 0
  Urine Urobilinogen ≥1 | 0 | 0 | 1 | 2
  Urine Bilirubin ≥1 | 0 | 0 | 1 | 0
  Urine Nitrite ≥1 | 0 | 0 | 1 | 0
  Urine Leukocytes ≥20: number analyzed (Participants) | 3 | 3 | 3 | 1
  Urine Leukocytes ≥20 | 0 | 1 | 1 | 0
  Urine Bacteria >20: number analyzed (Participants) | 3 | 3 | 3 | 1
  Urine Bacteria >20 | 0 | 1 | 0 | 0

6. Secondary Outcome: Number of Participants With Categorical Vital Signs Data
Description: Vital signs (systolic and diastolic blood pressure, and pulse rate) were obtained with participants after having sat calmly for at least 5 minutes.
Time Frame: Up to Day 4 (3 days after investigational product administration)
Population: All participants who received PF-06865571.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Systolic Blood Pressure (mmHg) Value <90 mmHg | 0 | 0 | 0 | 0
  Systolic Blood Pressure (mmHg) Change >=30 mmHg increase | 0 | 0 | 0 | 0
  Systolic Blood Pressure (mmHg) Change >=30 mmHg decrease | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) Value <50 mmHg | 0 | 0 | 1 | 1
  Diastolic Blood Pressure (mmHg) Change >=20 mmHg increase | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) Change >=20 mmHg decrease | 0 | 0 | 1 | 0
  Pulse Rate (beats per minute [bpm]) Value <40 bpm | 0 | 0 | 0 | 0
  Pulse Rate (bpm) Value >120 bpm | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Categorical Electrocardiogram (ECG)
Description: QT interval corrected using Fridericia's formula (QTcF) was obtained with participants. All scheduled ECGs were performed after the participant had rested quietly for at least 10 minutes in a supine position.
Time Frame: Up to Day 4 (3 days after investigational product administration)
Population: All participants who received PF-06865571.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  QTcF (millisecond [msec]) 450< Value <=480 | 0 | 0 | 1 | 1
  QTcF (msec) 480< Value <=500 | 0 | 0 | 0 | 0
  QTcF (msec) Value >500 | 0 | 0 | 0 | 0
  QTcF (msec) 30<= Change <=60 | 0 | 0 | 0 | 0
  QTcF (msec) Change >60 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 32 (31 days after investigational product administration)
Arm/Group | Cohort 1 (Without Hepatic Impairment) | Cohort 2 (Mild Hepatic Impairment) | Cohort 3 (Moderate Hepatic Impairment) | Cohort 4 (Severe Hepatic Impairment)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04091061/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-13): https://cdn.clinicaltrials.gov/large-docs/61/NCT04091061/SAP_001.pdf